CLINICAL TRIAL: NCT02580123
Title: Smile-Kids: Study on Complementary Feeding Transition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minho (Other)
Responsible Party: Principal Investigator, Helena Rafaela Vieira do Rosario, Dr, University of Minho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Smile-kids
Record Dates: First submitted 2015-04-13; First posted 2015-10-20 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Infant; Health Promotion; Nursery; Educators

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Experimental group (Experimental): Received the intervention program.
  Interventions: Behavioral: Intervention taught by trained educators
- Control group (No Intervention): received the standard care

INTERVENTIONS:
Behavioral: Intervention taught by trained educators
  Arms: Experimental group

SUMMARY:
The importance of families in the development of infants is well documented. Previous studies found that the prevalence of overweight and obesity is growing concerns in Portugal (Padez, Fernandes, Mourão, Moreira, & Rosado, 2004) and in the world (Ogden et al., 2014). More, there is evidence that habits acquired in early life might track into adulthood (Lien, Lytle, & Klepp, 2001; Lytle, Seifert, Greenstein, & McGovern, 2000; te Velde, Twisk, & Brug, 2007). Therefore, there is a need to lock overweight and obesity in early childhood in order to contribute to health gains during the entire life cycle. The main purpose of this research is to evaluate the impact of an intervention program based on parenting skills and feeding practices, on infant's growth, development and adherence to new foods in early infancy

Methods: 58 infants, 4-12 months from 25 nursery schools participated in this randomized trial and were randomly allocated to intervention and control group. Infant outcomes were performed at baseline and post-intervention and included anthropometry, dietary assessment and temperament. In addition maternal and family outcomes such as anxiety, dietary intake were also assessed at both times.

An intervention program was developed and Implemented according to two terms: educators' training with the researchers and the intervention with parents and infants developed by trained educators. The training program was developed between December 2013 and February 2014, according to the topics of healthy eating and nutrition and development of the infant. The control group received the standard care.

It is expected that this intervention program is able to promote healthy feeding practices to parents and nursery teachers. The results will be disseminated to the stakeholders and policymakers that work closely to the topic of this study. This will include papers' publication, participation in national and international meetings, contributing to the advance of research in this health area.

ELIGIBILITY:
Inclusion Criteria:

* Infants with 4-12 months

Exclusion Criteria:

* Infants with disability

Ages: 4 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2012-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Weight of the infant | 4 months up to 12 months of age
  Weight was measured with no clothes and no shoes, using standardized procedures,
Length of the infant | 4 months up to 12 months of age
  Length was measured according to standardized procedures.
Body Mass Index (BMI) of the infant | 4 months up to 12 months of age
  BMI was computed as the ratio weight/length2

SECONDARY OUTCOMES:
Dietary intake of infants | 4 months up to 12 months of age
  We used a questionnaires (2 day food record) to have data of dietary intake.
Temperament of the infant | 4 months up to 12 months of age
  Temperament was gathered with a questionnaire.
Family characteristics | 4 months up to 12 months of age
  Characteristics of infants´family, with a questionnaire about family income and dietary intake (Frequency Feeding Questionnaire)

REFERENCES:
- [Result] Padez C, Fernandes T, Mourao I, Moreira P, Rosado V. Prevalence of overweight and obesity in 7-9-year-old Portuguese children: trends in body mass index from 1970-2002. Am J Hum Biol. 2004 Nov-Dec;16(6):670-8. doi: 10.1002/ajhb.20080. PMID 15495229
- [Result] Ogden CL, Carroll MD, Flegal KM. Prevalence of obesity in the United States. JAMA. 2014 Jul;312(2):189-90. doi: 10.1001/jama.2014.6228. No abstract available. PMID 25005661
- [Result] Lien N, Lytle LA, Klepp KI. Stability in consumption of fruit, vegetables, and sugary foods in a cohort from age 14 to age 21. Prev Med. 2001 Sep;33(3):217-26. doi: 10.1006/pmed.2001.0874. PMID 11522162
- [Result] Lytle LA, Seifert S, Greenstein J, McGovern P. How do children's eating patterns and food choices change over time? Results from a cohort study. Am J Health Promot. 2000 Mar-Apr;14(4):222-8. doi: 10.4278/0890-1171-14.4.222. PMID 10915532
- [Result] te Velde SJ, Twisk JW, Brug J. Tracking of fruit and vegetable consumption from adolescence into adulthood and its longitudinal association with overweight. Br J Nutr. 2007 Aug;98(2):431-8. doi: 10.1017/S0007114507721451. Epub 2007 Apr 16. PMID 17433126